CLINICAL TRIAL: NCT00199615
Title: Follow-up of Patients With Curative-intent Surgical Resection for NSCLC : CT Scanning Versus 18 FDG Imaging.
Brief Title: Follow-up of Patients With Curative-intent Surgical Resection for NSCLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: I00021
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2005-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer, 18 FDG, PET
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PET — Intravenous injection of glucose labeled Fluor 18.Le patient remains fasted at least 6 hours before the start of the examination. The review lasted 1 hour, during which the patient should not move.

SUMMARY:
The guidelines and institutional practices recommended more frequent visits the two years following curative-intent therapy for non-small cell lung cancer (NSCLC).No international consensus is published concerning follow-up of resected NSCLC patients.Recent studies have outlined that positron emission tomography (PET) scanning may be accurate in early detection of recurrences by comparison to computed tomography (CT). The aim of this study is to compare follow-up by conventional methods versus PET. Patients are randomly assigned to two arms. In the first arm, thorax CT with liver and adrenal gland sections, abdominal ultrasonography and nuclear bone scintigraphy are performed every 6 months after surgery for two years. In the second arm, PET scanning is only. For brain metastasis detection, CT is performed in the two arms. Recurrences are detected during scheduled or unscheduled procedure in asymptomatic patients. PET and CT are interpreted separately by two nuclear physicians and two radiologists. The direct cost of follow-up procedure is determined in the two groups. The calculated sample is composed of 60 patients in each arm to detect significant difference. The Ethics Committee of Universitary Hospital of Limoges approves the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent resection for NSCLC
* Informed consent

Exclusion Criteria:

* Patients with a mixed histology profile that included small cell carcinoma or neuroendocrine tumor cells.
* Patients with non-resected NSCLC or with metastasis
* Patients who have previous malignancy, except basal cell carcinoma of the skin -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2001-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival from the date of operation to the date of recurrence or censured at the date of last follow-up visit or date of the death.

SECONDARY OUTCOMES:
- Overall survival from the date of the operation to the death
- Specificity, sensibility and accuracy of TEP to detect recurrence
- Direct cost of follow-up from the Frenc Healthcare insurance

CONTACTS AND LOCATIONS:
Overall Officials: Boris MELLONI, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Pathologie Respiratoire, Limoges, France

REFERENCES:
- [Background] Monteil J, Vergnenegre A, Bertin F, Dalmay F, Gaillard S, Bonnaud F, Melloni B. Randomized follow-up study of resected NSCLC patients: conventional versus 18F-DG coincidence imaging. Anticancer Res. 2010 Sep;30(9):3811-6. PMID 20944175